CLINICAL TRIAL: NCT04031690
Title: Health and Quality of Life Assessment Project for Caregivers of Idiopathic Pulmonary Fibrosis Patients
Acronym: HELP-IPF
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: BELTRAMO FRSR 2018
Record Dates: First submitted 2019-07-22; First posted 2019-07-24 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Idiopathic Pulmonary Fibrosis; Patient-caregiver Dyads
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patient-caregiver dyads
  Interventions: Other: Caregiver Quality of Life Questionnaires; Other: Patient Quality of Life Questionnaires

INTERVENTIONS:
Other: Caregiver Quality of Life Questionnaires — Measurement of quality of life at D0, M6 and M12 via SF-36, CarGOQoL and the one-dimensional Zarit score
Other: Patient Quality of Life Questionnaires — Quality of life measurement at D0, M6 and M12 via the SF-36

SUMMARY:
Idiopathic pulmonary fibrosis (IPF) is a chronic, disabling disease characterized by a progressive and irreversible deterioration in respiratory function, resulting in impaired quality of life (QoL) and patient dependence.

The factors involved in the alteration of QoL in these patients are the physical symptoms related to fibrosis (dyspnea, cough, fatigue) and psychological symptoms (anxiety and depression) as well as social, relational and financial factors, the experience of the disease and disability, the time required for diagnosis, the information received, and the initiation of a treatment such as oxygen therapy.

Caregivers primarily in chronic diseases (so-called natural or informal caregivers) provide partial or total assistance to a dependent person for activities of daily living for care, social support and maintenance of autonomy, administrative procedures, psychological support, communication, domestic activities or even financial assistance, often despite their own exhaustion and health issues.

Recent studies on the QoL of patient-caregiver dyads in IPF through semi-structured interviews highlight the role of previously identified factors in caregivers as well.

Investigators want to confirm the data obtained in a large population of patients and their caregivers in order to evaluate the QoL of caregivers and confirm the impact of its various factors on it in order to suggest ways to improve the lives of both the caregiver and the patient.

The hypothesis of investigators' work is that the QoL of caregivers of patients with IPF is altered, particularly by the patient's functional symptoms (cough, dyspnea, fatigue, anxiety and depression), the arrival of oxygen therapy in the home and the caregiver's social isolation.

Investigators believe that there are links and interactions between the caregiver's and patient's quality of life and therefore have an impact on the patient's care.

ELIGIBILITY:
Inclusion Criteria:

Patient inclusion criteria:

* Patient rescruited from prevalent cases and incidents of patients with IPF according to the diagnostic criteria of the 2011 ATS/ERS/JRS/ALAT recommendations, for which a follow-up is planned or is in progress
* Patient with a validated IPF diagnosis in multidisciplinary discussion in a Competence or Reference Centre. Regardless of the stage of the disease.
* Patient who has not opposed their enrollment in the study
* Adult patient
* Patient able to be assessed every 6 months by principal investigator
* A patient who can designate a non-professional primary caregiver regardless of kinship, age or involvement with the patient (the primary caregiver is defined as the person who works most frequently with the patient). Only one caregiver is retained per patient.
* Patient with no memory or comprehension problems and able to read and write French

Caregiver Inclusion Criteria:

* Caregiver designated by the patient as his or her primary caregiver
* Caregiver who has not opposed their participation in the study
* Adult caregiver
* Caregiver with no comprehension problems and able to read and write in French
* Caregiver with no memory problems

Exclusion Criteria:

* Person subject to a measure of legal protection (curatorship, guardianship)
* Person with a legal guardian
* Adult unable to consent

Patient non-inclusion criteria:

* Psychiatric, cognitive or neurological disorders making assessment impossible
* Patient suffering from another medical condition considered severe by the investigator and which may interfere with the consequences of IVF (for example, active cancers, motor disability of neurological origin, osteo-articular diseases inducing dependence...)
* Not likely to complete a self-administered questionnaire

Caregiver non-inclusion criteria:

* Psychiatric, cognitive or neurological disorders making assessment impossible
* Not likely to complete a self-administered questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consultation at the Reference or Competence Centre for Rare Adult Lung Diseases
Sampling Method: Non-Probability Sample
Enrollment: 151 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2020-09-28 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
The generic quality of life score SF-36 to measure caregivers' quality of life | Through study completion, an average of 12 months
  Measurement of caregivers' quality of life via the generic quality of life score SF-36 in each of the 8 dimensions of the component
The specific quality score CarGOQoL to measure caregivers' quality of life | Through study completion, an average of 12 months
  Measurement of caregivers' quality of life via the specific quality score CarGOQoL in each of the 10 dimensions of the component

SECONDARY OUTCOMES:
"subjective burden" of caregivers | Through study completion, an average of 12 months
  Measurement of the "subjective burden" of caregivers via the one-dimensional Zarit score
Patients' Quality of life | Through study completion, an average of 12 months
  Measurement of patients' quality of life via the generic quality of life score SF-36 in each of the 8 dimensions

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France